CLINICAL TRIAL: NCT05894967
Title: Moderators and Mediators of Perceptual Learning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020-0138; R01EY031226 (NIH); L&S/PSYCHOLOGY/PSYCHOLOGY (Other: UW Madison)
Record Dates: First submitted 2023-05-12; First posted 2023-06-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Change
Keywords: Vision Training

STUDY DESIGN:
Intervention Model Description: Participants in the younger adult cohort are randomized to 2 training conditions that they undergo sequentially (Arms C1-NCC). Participants in the older adult cohort are randomized to a single training condition (Arms OA1-OA5).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- C1 - Standard Perceptual Learning (SPL) (Experimental): Participants in younger cohort will complete SPL training during the first phase of training. In the cross-over they will then complete either SPL, LT, SS, MD, NT, TWF, or NCC.
  Interventions: Behavioral: C1 - Standard Perceptual Learning (SPL); Behavioral: C2 - Long Training (LT); Behavioral: C3 - Short Staircases (SS); Behavioral: C4 - Mixed Difficulty (MD); Behavioral: C5 - Noise Training (NT); Behavioral: C6 - Training with Flankers (TWF); Behavioral: No Contact Control
- C2 - Long Training (LT) (Experimental): Participants in younger cohort will complete LT training during the first phase of training. In the cross-over they will then complete either LT, SPL, or NCC.
  Interventions: Behavioral: C1 - Standard Perceptual Learning (SPL); Behavioral: C2 - Long Training (LT); Behavioral: No Contact Control
- C3 - Short Staircases (SS) (Experimental): Participants in younger cohort will complete SS training during the first phase of training. In the cross-over they will then complete either SS, SPL, or NCC.
  Interventions: Behavioral: C1 - Standard Perceptual Learning (SPL); Behavioral: C3 - Short Staircases (SS); Behavioral: No Contact Control
- C4 - Mixed Difficulty (MD) (Experimental): Participants in younger cohort will complete MD training during the first phase of training. In the cross-over they will then complete either MD, SPL, or NCC.
  Interventions: Behavioral: C1 - Standard Perceptual Learning (SPL); Behavioral: C4 - Mixed Difficulty (MD); Behavioral: No Contact Control
- C5 - Noise Training (NT) (Experimental): Participants in younger cohort will complete NT training during the first phase of training. In the cross-over they will then complete either NT, SPL, or NCC.
  Interventions: Behavioral: C1 - Standard Perceptual Learning (SPL); Behavioral: C5 - Noise Training (NT); Behavioral: No Contact Control
- C6 - Training with Flankers (TWF (Experimental): Participants in younger cohort will complete TWF training during the first phase of training. In the cross-over they will then complete eitherTWF, SPL, or NCC.
  Interventions: Behavioral: C1 - Standard Perceptual Learning (SPL); Behavioral: C6 - Training with Flankers (TWF); Behavioral: No Contact Control
- C7 - Parafoveal Training (PT) (Experimental): Participants in younger cohort will complete PT training during the first phase of training. In the cross-over they will then complete either PT, SV, CF, ExAT, EnAT, MF, or NCC.
  Interventions: Behavioral: C7 - Parafoveal Training (PT); Behavioral: C8 - Stimulus Variety (SV); Behavioral: C8a - Complex Features (CF); Behavioral: C9 - Exogenous Attention Training (ExAT); Behavioral: C10 - Endogenous Attention Training (EnAT); Behavioral: C11 - Multisensory Facilitation (MF); Behavioral: No Contact Control
- C8 - Stimulus Variety (SV) (Experimental): Participants in younger cohort will complete SV training during the first phase of training. In the cross-over they will then complete either SV, PT, or NCC.
  Interventions: Behavioral: C7 - Parafoveal Training (PT); Behavioral: C8 - Stimulus Variety (SV); Behavioral: No Contact Control
- C8a - Complex Features (CF) (Experimental): Participants in younger cohort will complete CF training during the first phase of training. In the cross-over they will then complete either CF, PT, NCC.
  Interventions: Behavioral: C7 - Parafoveal Training (PT); Behavioral: C8a - Complex Features (CF); Behavioral: No Contact Control
- C9 - Exogenous Attention Training (ExAT) (Experimental): Participants in younger cohort will complete ExAT training during the first phase of training. In the cross-over they will then complete either ExAT, PT, NCC.
  Interventions: Behavioral: C7 - Parafoveal Training (PT); Behavioral: C9 - Exogenous Attention Training (ExAT); Behavioral: No Contact Control
- C10 - Endogenous Attention Training (EnAT) (Experimental): Participants in younger cohort will complete EnAT training during the first phase of training. In the cross-over they will then complete either EnAT, PT, NCC.
  Interventions: Behavioral: C7 - Parafoveal Training (PT); Behavioral: C10 - Endogenous Attention Training (EnAT); Behavioral: No Contact Control
- C11 - Multisensory Facilitation (MF) (Experimental): Participants in younger cohort will complete MF training during the first phase of training. In the cross-over they will then complete either MF, PT, NCC.
  Interventions: Behavioral: C7 - Parafoveal Training (PT); Behavioral: C11 - Multisensory Facilitation (MF); Behavioral: No Contact Control
- No Contact Control (Other): Participants in younger cohort will complete NCC training during the first phase of training. In the cross-over they will then complete either SPL, LT, SS, MD, NT, TWF, PT, SV, CF, ExAT, EnAT, MF, NCC.
  Interventions: Behavioral: C1 - Standard Perceptual Learning (SPL); Behavioral: C2 - Long Training (LT); Behavioral: C3 - Short Staircases (SS); Behavioral: C4 - Mixed Difficulty (MD); Behavioral: C5 - Noise Training (NT); Behavioral: C6 - Training with Flankers (TWF); Behavioral: C7 - Parafoveal Training (PT); Behavioral: C8 - Stimulus Variety (SV); Behavioral: C8a - Complex Features (CF); Behavioral: C9 - Exogenous Attention Training (ExAT); Behavioral: C10 - Endogenous Attention Training (EnAT); Behavioral: C11 - Multisensory Facilitation (MF); Behavioral: No Contact Control
- OA1 - Standard Perceptual Learning (Experimental): Participants in older cohort will complete SPL condition.
  Interventions: Behavioral: C1 - Standard Perceptual Learning (SPL)
- OA2 - Noise Training (Experimental): Participants in older cohort will complete NT condition.
  Interventions: Behavioral: C5 - Noise Training (NT)
- OA3 - Training with Flankers (Experimental): Participants in older cohort will complete TWF condition.
  Interventions: Behavioral: C6 - Training with Flankers (TWF)
- OA4 - Stimulus Variety (Experimental): Participants in older cohort will complete SV condition.
  Interventions: Behavioral: C8 - Stimulus Variety (SV)
- OA5 - No Contact Control (Experimental): Participants in older cohort will complete NCC condition.
  Interventions: Behavioral: No Contact Control

INTERVENTIONS:
Behavioral: C1 - Standard Perceptual Learning (SPL) — Each trial starts with a fixation point (500ms) after which a Gabor (1° radius, at cut-off SF of 25% accuracy, estimated from Pre-Test CSF, at either 45° or 135°) appears for 128ms. The task is to indicate whether the Gabor was tilted left or right. Gabor contrast will be controlled by a 3/1 staircase (converging on approximately ~80% contrast threshold) across all training sessions.
  Arms: C1 - Standard Perceptual Learning (SPL); C2 - Long Training (LT); C3 - Short Staircases (SS); C4 - Mixed Difficulty (MD); C5 - Noise Training (NT); C6 - Training with Flankers (TWF; No Contact Control; OA1 - Standard Perceptual Learning
Behavioral: C2 - Long Training (LT) — Will be the same as the SPL with the exception that each session in LT will be twice as long as in SPL.
  Arms: C1 - Standard Perceptual Learning (SPL); C2 - Long Training (LT); No Contact Control
Behavioral: C3 - Short Staircases (SS) — Will be largely the same as SPL with the only difference being a change to the adaptive procedure. SS will use so-called "short-staircases," which are initialized at 60% contrast with steps of .05 log units and employs a 3/1 staircase that after every 40 trials is reset (the "short" in "short-staircases") back to 60% contrast.
  Arms: C1 - Standard Perceptual Learning (SPL); C3 - Short Staircases (SS); No Contact Control
Behavioral: C4 - Mixed Difficulty (MD) — This condition will be identical to SPL with the exception that two staircases - one a 2/1 staircase producing difficulties centered around 60-70% accuracy, the other a 4/1 staircase producing difficulties centered around 85-95% accuracy - will be utilized to control the stimuli.
  Arms: C1 - Standard Perceptual Learning (SPL); C4 - Mixed Difficulty (MD); No Contact Control
Behavioral: C5 - Noise Training (NT) — The NT condition will be the same as SPL with the exception that contrast thresholds will be estimated in 5-different levels of external noise (10%, 15%, 20%, 25%, 30%).
  Arms: C1 - Standard Perceptual Learning (SPL); C5 - Noise Training (NT); No Contact Control; OA2 - Noise Training
Behavioral: C6 - Training with Flankers (TWF) — TWF will be reasonably different from the standard SPL task. Here, on 50% of trials a target Gabor will be presented at either 45° or 135° (as in SPL) and will be flanked by two collinear Gabors. On the remaining 50% of trials, flankers will be present without a target. TWF is thus a yes/no detection task, which is necessary since the collinear flankers fully indicate the target orientation. In different 20-trial mini-blocks the flankers will appear either lambda, 1.5 lambda, or 2 lambda from the target (i.e., closer or further from the target) and target contrast will be controlled by a 3/1 staircase separately for each spacing.
  Arms: C1 - Standard Perceptual Learning (SPL); C6 - Training with Flankers (TWF; No Contact Control; OA3 - Training with Flankers
Behavioral: C7 - Parafoveal Training (PT) — The PT condition is the baseline for C8-C11 (all of which involve parafoveally presented targets). In PT, we utilize the same task as in SPL, however, in PT, in addition to central training, targets will also appear in one of two peripheral locations (5° eccentricity; angles = 135° and 270°). The location of targets will be randomized trial-wise so as to discourage eye-movements and independent 3/1 staircases will be run at each location. By training only 2 peripheral locations we can measure the extent to which training gives rise to location transfer (e.g., in transfer tasks examining performance at 8 different locations - 2 trained locations and 6 untrained locations). Furthermore, training at the central location facilitates comparisons between PT and SPL.
  Arms: C10 - Endogenous Attention Training (EnAT); C11 - Multisensory Facilitation (MF); C7 - Parafoveal Training (PT); C8 - Stimulus Variety (SV); C8a - Complex Features (CF); C9 - Exogenous Attention Training (ExAT); No Contact Control
Behavioral: C8 - Stimulus Variety (SV) — The base task for SV is the PT condition. However, SV employ 20 trial mini-blocks of different SFs (.75, 1.5, 3, 6, 12, 24 cpd) and locations (45°, 135°, 225°, 315° - i.e., more locations than PT, but not the full set tested in the transfer battery) with separate staircases for each SF and location. Orientations will also be drawn from a larger set (22.5°, 45°, 67.5° - for which participants respond "clockwise" and 112.5°, 135°, 157.5° - for which participants respond "counter-clockwise") and will vary on a trial-by-trial basis. This design holds-out 4 locations and 2 orientations to address transfer.
  Arms: C7 - Parafoveal Training (PT); C8 - Stimulus Variety (SV); No Contact Control; OA4 - Stimulus Variety
Behavioral: C8a - Complex Features (CF) — This is the same as C8, however we will use band-pass filtered stimuli similar to what has been done by a number of groups including Hussein et al.
  Arms: C7 - Parafoveal Training (PT); C8a - Complex Features (CF); No Contact Control
Behavioral: C9 - Exogenous Attention Training (ExAT) — Stimuli will be presented in a similar manner as in PT. However, in ExAT, a 100% valid cue, a small black dot - 48ms duration with an 96ms SOA prior to stimulus onset - will appear above the target location on each trial.
  Arms: C7 - Parafoveal Training (PT); C9 - Exogenous Attention Training (ExAT); No Contact Control
Behavioral: C10 - Endogenous Attention Training (EnAT) — Stimuli will be presented in a similar manner as in PT. However, in EnAT, a 100% valid cue (letter UL, LR; standing for upper left and lower right, respectively) - 150ms duration with an 500ms SOA prior to stimulus onset - will appear at the fixation point.
  Arms: C10 - Endogenous Attention Training (EnAT); C7 - Parafoveal Training (PT); No Contact Control
Behavioral: C11 - Multisensory Facilitation (MF) — MF utilizes the same basic task structure as in ExEAT, however, rather than a visual cue, an auditory cue will be used (50ms, 1000hz tone with sound location determined by convolving sound with generic head-related transfer function, kemar large ears.
  Arms: C11 - Multisensory Facilitation (MF); C7 - Parafoveal Training (PT); No Contact Control
Behavioral: No Contact Control — While not a "training condition" one type of experience that could be part of a condition is a no contact control (i.e., where participants do no training activities over the same rough time span as for the other training tasks).
  Arms: C1 - Standard Perceptual Learning (SPL); C10 - Endogenous Attention Training (EnAT); C11 - Multisensory Facilitation (MF); C2 - Long Training (LT); C3 - Short Staircases (SS); C4 - Mixed Difficulty (MD); C5 - Noise Training (NT); C6 - Training with Flankers (TWF; C7 - Parafoveal Training (PT); C8 - Stimulus Variety (SV); C8a - Complex Features (CF); C9 - Exogenous Attention Training (ExAT); No Contact Control; OA5 - No Contact Control

SUMMARY:
This is a research study about how training can impact performance on cognitive tasks. Participants are between 18 and 30 and 60 to 85 years of age, have normal (or corrected to normal) vision, and have no neurological conditions that would preclude their ability to complete computerized cognitive tasks. Up to 1140 participants will be on study for up to 8 weeks.

DETAILED DESCRIPTION:
This study addresses the fundamental issue of specificity and generality of training in the context of Perceptual Learning (PL). PL broadly encompasses the set of mechanisms through which experience with the environment gives rise to changes in perceptual processing. Careful research in this domain can greatly enhance basic understanding of the perceptual systems and the plasticity of these systems. Furthermore, translational approaches underpinned by the basic science of PL are becoming increasingly prominent. This includes a host of emerging translational approaches for the rehabilitation of both perceptual deficits and for cognitive training, which are believed to share cortical plasticity mechanisms. However, while existing research provides evidence that PL approaches can improve perceptual skills, the ability to develop effective interventions is limited by a lack of understanding of the behavioral outcomes associated with different PL approaches. One major obstacle to successful translation of PL is that the field to-date has been strongly driven by "novel" and "provocative" findings demonstrated via small N studies with very few projects digging deep to achieve robust and reliable results. In turn, not surprisingly, the field of PL, like many others in psychology, has suffered from numerous replication challenges. Here the investigators address these limitations by comparing a large number of different training tasks using common outcome measures and in a large subject population. Each training tasks involves a different "critical feature" for learning proposed by one or more research groups. However, these training tasks have never been directly compared or contrasted. Robust and reliable results will be achieved by training a large sample of participants on PL tasks and assess the outcomes via a common set of measures. The investigators will also collect a broad assessment of individual differences, which will provide a unique dataset that can resolve controversies in the literature and lead to new understandings. The proposed analytical approach tests several key hypotheses in the field, explores the extent to which different training approaches lead to systematically different profiles of learning, and examines how these can differ based upon the individuals being trained.

The present study investigates the mechanisms of Perceptual Learning (PL), with a focus on training task characteristics that induce generalizable enhancements in visual performance (i.e., that produce benefits on tasks beyond just the trained task, as this is critical for training to have translational value). To achieve this, the investigators target PL of spatial vision in human subjects, which is the most common target of PL in basic science research.

The investigators run a large number of participants across 12 separate conditions thought to mediate effects of PL (e.g., training with flanking stimuli, use of noise, manipulating difficulty during training, multisensory facilitation with sound, training with a diversity of stimuli, and cueing attention during training) using common outcome measures, and analyze both the effect of training condition and individual differences that impact learning. A novel crossover design is used to train participants in the younger cohort sequentially on two tasks and examine learning and generalization to determine which methods involve redundant or independent processes. It is noted that the first phase of training is the primary clinical trial and that the crossover is to address a mechanistic question regarding interactions of different training types. It is hypothesized that training with mostly difficult, precise stimuli will give rise to less generalization than training with easy, imprecise stimuli after sequential double training.

The investigators also specifically examine biological variables, such as sex and age, in addition to personality traits, sleep habits, motivation, and individual differences in baseline performance to gain a more complete understanding of how these factors may moderate outcomes of PL (including generalization to more real-world contexts, such as reading). It is hypothesized that a number of individual differences, both cognitive and personality based, will predict PL outcomes.

Participants in the younger cohort will be randomized to 1 of 12 arms, with each arm consisting of two conditions (of twelve possible conditions) that participants undergo sequentially. Participants in the older adult cohort will be randomized to 1 of 5 arms, with each arm consisting of a single condition.

ELIGIBILITY:
Inclusion Criteria:

* between18 and 30 years of age (younger cohort)
* between 60 and 85 years of age (older cohort)
* Corrected vision of 20/40 or better (as assessed with an eye chart)
* No reported incidence of retinal pathology or neurological disease

Exclusion Criteria:

* Corrected vision of 20/40 or worse
* Evidence of retinal pathology or retinal disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1140 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Near Transfer Task | Baseline to Post-test 2, an average of 5-8 weeks
  We will utilize an overarching task structure that allows us to assess learning on trained stimuli and transfer to untrained stimuli; locations, orientations, stimulus timings (e.g., we will assess contrast sensitivity for 6 different orientations). A trial begins with a fixation-point presented for 500ms. A target stimulus then appears for 128ms and then disappears (this timing was chosen to preclude participants making eye-movements to the stimuli). The participant is then required to respond by indicating the orientation of the stimulus (e.g., the major axis of a Gabor stimulus or gap-side of a C stimulus). In contrast tests, a staircase is run on the contrast of the target stimulus. In acuity tests, a staircase is run on the size of the stimulus. In parafoveal tests, stimuli are presented at 5° eccentricity.
Change in Transfer to Visual Search | Baseline to Post-test 2, an average of 5-8 weeks
  In a T/L annular visual-search task (1° stimuli, presented at 5° eccentricity at each of 8 evenly spaced locations), on each trial, 7 positions are filled with a distractor (upside-down Ls, half black and half white), while 1 position contains a target (rightside-up T that is either white or black). Stimuli are presented for 256ms and, after a variable SOA, a stimulus-mask (asterixis) appears. Participants report the color of the T. A 3/1 staircase controls the SOA of the mask (shorter SOAs = less time between stimulus and mask = more difficult). This task tests how training impacts processing time (i.e., time necessary to find and identify targets). Also, given that the same locations are used as in the parafoveal training, we can also estimate the extent to which transfer to visual search occurs and, if so, whether it is specific to the trained location.
Change in Transfer to Reading | Baseline to Post-test 2, an average of 5-8 weeks
  To understand visual performance related to reading, we employ the MNRead task, where participants read short sentences out-loud at various font-sizes. Dependent variables include reading speed, minimal text-size (another measure of acuity), and also critical print-size (text-size at which reading speed slows down).
Change in Transfer to Auditory Attention | Baseline to Post-test 2, an average of 5-8 weeks
  The procedure is based upon a speaker-on-speaker task where participants choose between 36 call signs (a color and number) spoken by a speaker. This task measures auditory thresholds for speech in the presence of other talkers, when all talkers are spatially collocated compared to when they are spatially offset.

CONTACTS AND LOCATIONS:
Overall Officials: C. Shawn Green, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - University of California, Riverside, California
  - Northeastern University, Boston, Massachusetts
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No